CLINICAL TRIAL: NCT04295317
Title: Eﬀect of PD-1 Antibody (SHR-1210) Combined with Capecitabine Treatment After Resection of Intrahepatic Cholangiocarcinoma with High Risk of Recurrence : a Phase 2 Study.
Brief Title: PD-1 Antibody (SHR-1210) Plus Capecitabine in Patients with Intrahepatic Cholangiocarcinoma After Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhou, professor, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2019-276(2)R
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: PD-1 Antibody; Capecitabine; Intrahepatic Cholangiocarcinoma; Adjuvant therapy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined the therapy using Capecitabine and PD-1 (Experimental): PD1 antibody SHR-1210 D1 200 mg every three weeks; Three weeks is a course of treatment with a total of 8 courses, or the patient has tumor recurrence or metastasis (requires imaging to determine tumor recurrence or metastasis) Capecitabine 2500mg / m2, 2 times/d for 2 weeks, followed by 1 week of stopping ,Three weeks is a course of treatment with a total of 8 courses, or the patient has tumor recurrence or metastasis (requires imaging to determine tumor recurrence or metastasis)
  Interventions: Drug: PD-1 blocking antibody SHR-1210; Drug: Capecitabine

INTERVENTIONS:
Drug: PD-1 blocking antibody SHR-1210 — PD1 antibody SHR-1210 D1 200 mg every three weeks; Three weeks is a course of treatment with a total of 8 courses, or the patient has tumor recurrence or metastasis (requires imaging to determine tumor recurrence or metastasis)
Drug: Capecitabine — Capecitabine 2500mg / m2/ d, 2 times/d for 2 weeks, followed by 1 week of stopping ,Three weeks is a course of treatment with a total of 8 courses, or the patient has tumor recurrence or metastasis (requires imaging to determine tumor recurrence or metastasis)

SUMMARY:
SHR-1210 is a humanized anti-PD-1 Immunoglobulin G4 (IgG4) monoclonal antibody. This is an open- label,single center,non-randomized ,single arm exploratory study . This clinical study is an investigator-initiated clinical trial(IIT) .The objective of this study is to evaluate the efficacy and safety of therapy with anti-PD-1 antibody SHR-1210 plus Capecitabine in patients with Intrahepatic Cholangiocarcinoma After Surgery.

ELIGIBILITY:
Inclusion Criteria:

* age:18-75 years, male or femal;
* Intrahepatic Cholangiocarcinoma confirmed by histopathology, R0 resection was classified as Stage IB, Stage II, Stage IIIA, Stage IIIB, or Stage IA with histolgoic grade G3 according to AJCC TNM (8th edition, 2017);
* No extrahepatic metastases;
* preoperative assessment of Child-Pugh A，ECOG Performance Status 0-1;
* Subjects with chronic HBV infection must have HBV-DNA <500 IU / ml;
* Functional indicators of vital organs meet the following requirements: Neutrophils ≥1.5*109/L; platelets≥50*109/L; hemoglobin≥90g/l; Alanine aminotransferase （ALT） and Aspartate aminotransferase （AST） ≤ 2.5 times ULN,total bilirubin≤1.5 ULN; International standardized ratio (INR) ≤2.3ULN,creatinine ≤1.5 ULN;
* No tumor recurrence or metastasis was observed.

Exclusion Criteria:

* Pathological diagnosis of hepatocellular carcinoma, mixed liver cancer, hilar bile duct cancer;
* No anti-tumor treatment for Intrahepatic Cholangiocarcinoma, including chemotherapy and topical treatment, before surgery;
* Known history of hypersensitivity to macromolecular protein preparation or any components of the SHR- 1210 formulation;
* Tumors are not completely removed, or postoperative pathology suggests non-Intrahepatic Cholangiocarcinoma or other malignant components;
* Subjects with any active autoimmune disease or history of autoimmune disease;
* Uncontrolled clinically significant heart disease, including but not limited to the following: (1) > NYHA II congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention;
* Active infection or an unexplained fever > 38.5°C during screening or before the first scheduled day of dosing (subjects with tumor fever may be enrolled at the discretion of the investigator);
* Received a live vaccine within 4 weeks of the first dose of study medication;
* .Pregnancy or breast feeding;
* Decision of unsuitableness by principal investigator or physician-in- charge.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival | 24 months
  From the date of enrollment to the date of diagnosis of tumor recurrence

SECONDARY OUTCOMES:
overall survival | 24 months
  From the date of enrollment to the date of death
the potential side effects | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, professor, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Z, Li L, Huang P, Tu H, Zhang X, Yu L, Liang F, Huang C, Qiu S, Ye Q, Ding Z, Huang X, Shi Y, Song K, Sun H, Wang X, Xu Y, Yu Y, Gao Q, Zhang L, Fan J, Zhou J. Adjuvant camrelizumab combined with capecitabine in patients with intrahepatic cholangiocarcinoma after surgical resection in China (ACC): a single-arm, single-centre, open-label, phase 2 trial. Lancet Gastroenterol Hepatol. 2026 Feb;11(2):124-136. doi: 10.1016/S2468-1253(25)00268-7. Epub 2025 Nov 27. PMID 41319673